CLINICAL TRIAL: NCT04783337
Title: Local Remodelling and Mechanoregulation of Bone Fracture Healing in Healthy, Aged, and Osteoporotic Humans
Brief Title: Local Remodelling of Bone Fracture Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Collaborators: ETH Zurich (Other); University Hospital Ulm (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: I-3258-B27_microCT Radius
Record Dates: First submitted 2021-02-15; First posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-02

CONDITIONS: Fracture Healing; Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HR-pQCT (high resolution computertomograph) (Experimental): This arm is the inverventional group for all collected cases. No other arms are available as comparator or control. All patients are treated the same.
  Description of the intervention in the section "Intervention".
  Interventions: Diagnostic Test: HR-pQCT (high resolution computertomograph); Diagnostic Test: Blood withdrawal

INTERVENTIONS:
Diagnostic Test: HR-pQCT (high resolution computertomograph) — In addition to determining the bone density, a quantitative bone structure analysis with measurement of the number of thickness and distribution of the trabeculae can also be carried out. In addition, the finite element analysis (FEA) allows strength models of the examined bone to be created from the data of the hr-pqCTs. In this way, the osseous consolidation of the fracture can not only be observed, but also tested for resilience with the help of mathematical models.
Diagnostic Test: Blood withdrawal — Bone remodeling blood marker: S-CTX (Crosslaps), S-TRA5b ( tartrate-resistant acid phosphatase), S-PINP (Procollagen type 1 amino-terminal propeptide), BALP, Calcium, parathyroid hormone, 25-OH-Vitamin D3 (HPLC)

SUMMARY:
The aim of our study is to improve a mathematical model (FAE) of human bone healing using the example of the distal spoke fracture. Computer-aided strength analyzes of data from hr-pqCTs should provide information about the fracture strength and quality of the newly formed bone at defined times. Laboratory parameters from sober blood analyzes, bone remodeling markers, competitive x-rays, the course of pain, range of motion, grip strength and other easily accessible parameters should be evaluated with the above-mentioned analyzes.

DETAILED DESCRIPTION:
So far, empirical values have mainly been used to assess fracture healing. The clinical parameter used is freedom from pain over the fracture, and native radiology the callus formation. In the case of anatomically reduced fractures, however, this can hardly be observed. In the case of a distal radius fracture, it is assumed that the total time to complete healing and resilience is one year. However, this has not been proven biomechanically.

The high-resolution peripheral quantitative computed tomography offers the possibility of precisely describing the healing process in the high-resolution range using the trabecular structure, bone density, bone volume and tissue composition. The finite element analysis can then be used to calculate the load-bearing capacity of the bone and to create failure models. The distal radius fracture is one of the most common fractures in humans, especially in osteoporosis. Due to its frequency and easily accessible fracture localization, it is an ideal model for investigating fracture healing. The additional examination of blood and urine for bone loss markers can provide further information on the healing process in conjunction with the image data.

It is a prospective cohort study. The collected data are compared on the one hand with preliminary examinations of the injured side in the sense of creating a model and on the other hand with the healthy, non-fractured side in order to compare the strength of the fracture.

Performing the X-ray and HR-pQCTs leads to radiation exposure which, however, can be classified as low. (X-ray: 0.02 mSv / image; HR-pQCT: between 0.003 - 0.006 mSv / stack image). The DXA examination on the distal radius, femur / hip + lumbar spine requires 0.405 mSv. With 18 x-rays and 24 HR-pQCTs and 1 DXA per patient, there is a radiation exposure of 0.837 - 0.909 mSv over the course of the academic year.

Blood will also be taken and urine samples will be collected. Together with the clinical examination and filling in the questionnaire, each examination should take approx. 45 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Conservatively treated distal radius fracture
* Able and agree to sign a written consent
* Able and agree to attend the follow-up examinations
* Able to understand the national language both in writing and orally to a minimum

Exclusion Criteria:

* Age under 18
* Comminuted fracture
* Bilateral spoke fracture
* unstable fracture with indication for surgical treatment
* open spoke fracture
* Adjacent fractures or injuries
* Previous injury to the distal radius
* The patient cannot give consent due to physical or mental disabilities
* Patient is not available for regular check-ups (abroad)
* The patient does not have full legal capacity
* Alcohol and drug abuse
* Current treatment with steroids
* Multiple trauma
* Illnesses or disorders that restrict the movement of a hand (apoplexy, hemiparesis, neuromuscular or rheumatic disease, severe mental or metabolic diseases)
* Rheumatoid arthritis
* Previous radio or chemotherapy within the last year
* Currently participating in a pharmaceutical study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2015-12-10 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Strength analysis of the distal radius fracture | 1 year
  The aim of our study is to create a mathematical model of human bone healing using the example of a distal radius fracture. Computer-aided strength analyzes of data from hr-pqCTs should provide information about the fracture strength and quality of the newly formed bone at defined times.(finite element analysis- FEA)

SECONDARY OUTCOMES:
Rate of bone density | 1year
  Amount of bone mineral in bone tissue, using DXA Scan (Dual-xray absorbtiometry).
Bone remodeling markers (blood analysis) | 1year
  Concentration of bone remodeling markers of (sober) blood samples with signs of healing in hr-pqCT and conventional X-rays. Blood markers of bone remodeling are: S-CTX (Crosslaps), S-TRA5b ( tartrate-resistant acid phosphatase), S-PINP (Procollagen type 1 amino-terminal propeptide), BALP, Calcium, parathyroid hormone, 25-OH-Vitamin D3 (HPLC).
  Increaseing bone turnover values during healing period.
Patient Reported Outcome (function) | 1 year
  Percentage of the patients with reduced or normal outcome after fractures using questionnaires like the Michigan Wrist Score in correlation of the healing process. This is a score reporting the functional outcome, satisfaction and quality of life. Best score is 100%, least score 0%.
Patient Reported Outcome (pain) | 1 year
  Percentage of the patients with remaining pain after fracture using the visual analog scale in correlation of the healing process. The scale reports about the intensity of pain. The maximum pain and least score is 10, and the best score is 0 which means "no pain".
Clinical outcome (range of motion) | 1 year
  Degree of the possible range of motion using a goniometer to measure the movement angles in correlation of the healing process. The better the range of motion the higher the value. Normally the following limits are given:
  Radial: least 0 degree, maximum: 20 degree Ulnar: least 0 degree, maximum: 40 degree Extension: least 0 degree, maximum: 70 degree Flexion: least 0 degree, maximum: 70 degree Pronation: least 0 degree, maximum: 90 degree Supination: least 0 degree, maximum: 90 degree
Clinical outcome (grip strength wrist) | 1 year
  Extent of possible grip strength measurement using dynanometer in correlation of the healing process.
  Minimum: 0 kilogram Maximum: 80 kg

IPD SHARING:
Plan to Share IPD: No